CLINICAL TRIAL: NCT01531595
Title: Phase 2 Study of Bevacizumab in Combination with Alternating XELIRI and XELOX As First-line Treatment of Patients with Metastatic Colorectal Cancer
Brief Title: Study of Bevacizumab in Combination with Alternating XELIRI and XELOX in Metastatic Colorectal Cancer
Acronym: AXOAXI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pia Osterlund (Other)
Responsible Party: Sponsor-Investigator, Pia Osterlund, Principal Investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-003137-33
Record Dates: First submitted 2012-02-03; First posted 2012-02-13 (Estimated); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Irinotecan; Oxaliplatin; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy plus bevacizumab (Experimental): Bevacizumab plus alternating XELOX x3 cycles (capecitabine + oxaliplatin) and XELIRI x3 cycles (capecitabine + irinotecan)
  Interventions: Drug: Bevacizumab plus alternating XELOX/XELIRI

INTERVENTIONS:
Drug: Bevacizumab plus alternating XELOX/XELIRI — 3 cycles of XELOX+bevacizumab alternating with 3 cycles XELIRI+bevacizumab until disease progression
  Other Names: Avastin (bevacizumab); Xeloda (capecitabine); irinotecan; oxaliplatin; XELIRI (capecitabine + irinotecan); XELOX (capecitabine + oxaliplatin)

SUMMARY:
* Open-label, single-arm, phase II study of bevacizumab (AvastinTM) in combination with alternating XELIRI (capecitabine+irinotecan) and XELOX (capecitabine+oxaliplatin) as first-line treatment of patients with metastatic colorectal cancer.
* Primary objective: Progression Free Survival (PFS),
* To assess overall resectability in patients with metastatic colorectal cancer, postoperative morbidity and outcomes after resection.
* Secondary objectives: To assess response rates according to RECIST criteria, failure free survival (TTF) and overall survival (OS), Quality of life according to 15-dimensional instrument (15D) questionnaire, To radiologically assess tumour density and morphology, and assess alternative radiologic response evaluation in comparison with RECIST response criteria, Biomarker evaluation to measure plasma biomarkers, tumour blocks and DNA polymorphisms that may predict drug effects, safety, resectability and clinical behaviour of the tumour

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed diagnosis of colorectal cancer (CRC), chemotherapy naïve for metastatic disease (prior adjuvant chemotherapy more than 6 months previously for CRC allowed), who are scheduled to start first line chemotherapy for metastatic disease
2. Age > 18
3. Measurable or evaluable metastatic disease
4. Performance status Eastern co-operative oncology group (ECOG) performance status 0-2
5. Life expectancy greater than 3 months
6. Normal Thrombocytes, neutrophils, Aspartate amino transferase/Alanine amino transferase, Alkaline phosphatase, Serum bilirubin, Serum Creatinine, Urine dipstick of proteinuria.
7. Women of childbearing potential must have a negative serum pregnancy test done prior to the administration of bevacizumab. Patient and their partner should have adequate contraception up to at least 6 months after last treatment completion or the last drug dose, whatever happens first
8. Signed written informed consent according to international council for harmonization (ICH)/Good clinical practice (GCP) and the local regulations (approved by the Independent Ethics Committee (IEC)) will be obtained prior to any study specific screening procedures
9. Patient must be able to comply with the protocol

Exclusion Criteria:

1. Prior treatment with first-line chemotherapy for metastatic CRC
2. Adjuvant treatment within 6 months
3. Major surgical procedure (placing of central venous access device and liver biopsy etc are considered minor procedure), open biopsy or significant traumatic injury within 28 days prior to Day 0 (Patients must have recovered from any major surgery)
4. Near future planned radiotherapy for underlying disease (prior completed radiotherapy treatment allowed)
5. Clinical or radiological evidence of central nervous system (CNS) metastases
6. Past or current history within the last 2 years of malignancies except for the indication under this study and curatively treated basal and squamous cell carcinoma of the skin or in-situ carcinoma of the cervix
7. Serious non-healing wound or ulcer
8. Evidence of bleeding diathesis or coagulopathy
9. Uncontrolled hypertension
10. Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤ 6 months), myocardial infarction (≤ 6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
11. Treatment with any investigational drug within 30 days prior to enrolment
12. Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the treatment or patient at high risk from treatment complications
13. Chronic daily intake of aspirin (> 325 mg/day) or clopidogrel (> 75 mg/day)
14. Pregnancy (positive serum pregnancy test) and lactation
15. Any other serious or uncontrolled illness which, in the opinion of the investigator, makes it undesirable for the patient to enter the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Resectability of metastases | 5 years
  To evaluate technical resectability rate of colorectal cancer metastasis after conversion therapy
Efficacy of alternating therapy | 5 years
  Progression free survival rate at 12 months

SECONDARY OUTCOMES:
Response of alternating therapy | 5 years
  To assess response rates according to RECIST criteria
Efficacy of treatment | 5 years
  Overall survival
Progression-free survival | 5 years
  Progression-free survival
Translational research | 10 years
  Prognostic and predictive factors

CONTACTS AND LOCATIONS:
Overall Officials: Pia Osterlund, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Department of Oncology, Helsinki, Finland